CLINICAL TRIAL: NCT01376323
Title: A Multicenter, Two Part, Randomized, Parallel Group, Placebo and Sitagliptin Controlled Study to Evaluate the Safety and Efficacy of GSK256073 Administered Once or Twice Daily for 12 Weeks in Subjects With Type 2 Diabetes Mellitus Who Are Being Treated With Metformin
Brief Title: A Study of GSK256073 in Subjects With Type 2 Diabetes Mellitus Who Are Being Treated With Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114728
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Results first posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Safety; Dose Ranging; Efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 8-chloro-3-pentyl-1H-purine-2,6(3H,7H)-dione; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- GSK256073 1mg bid (Experimental): GSK256073 1mg capsule taken orally twice a day
  Interventions: Drug: GSK256073 1mg
- GSK256073 2mg qd (Experimental): GSK256073 2 x 1mg capsule taken orally once a day
  Interventions: Drug: GSK256073 1mg
- GSK256073 5mg bid (Experimental): GSK256073 5mg capsule taken orally twice a day
  Interventions: Drug: GSK256073 5mg
- GSK256073 10mg qd (Experimental): GSK256073 2 x 5mg capsule taken orally once a day
  Interventions: Drug: GSK256073 5mg
- GSK256073 10mg bid (Experimental): GSK256073 10mg capsule taken orally twice a day
  Interventions: Drug: GSK256073 10mg
- GSK256073 20mg qd (Experimental): GSK256073 2x 10mg capsule taken orally once a day
  Interventions: Drug: GSK256073 10mg
- GSK256073 25mg bid (Experimental): GSK256073 25mg capsule taken orally twice a day
  Interventions: Drug: GSK256073 25mg
- GSK256073 50mg qd (Experimental): GSK256073 2x 25mg capsule taken orally once a day
  Interventions: Drug: GSK256073 25mg
- Placebo (Placebo Comparator): Matching placebo capsules taken orally either once a day or twice a day
  Interventions: Drug: Placebo
- Sitagliptin 100mg qd (Active Comparator): Commercially available Sitagliptin 100mg capsules taken once a day
  Interventions: Drug: Sitagliptin 100mg

INTERVENTIONS:
Drug: GSK256073 1mg — GSK256073 1mg capsule
  Arms: GSK256073 1mg bid; GSK256073 2mg qd
Drug: GSK256073 5mg — GSK256073 5mg capsule
  Arms: GSK256073 10mg qd; GSK256073 5mg bid
Drug: GSK256073 10mg — GSK256073 10mg capsule
  Arms: GSK256073 10mg bid; GSK256073 20mg qd
Drug: GSK256073 25mg — GSK256073 25mg capsule
  Arms: GSK256073 25mg bid; GSK256073 50mg qd
Drug: Placebo — placebo capsule
  Arms: Placebo
Drug: Sitagliptin 100mg — Sitagliptin 100mg capsule
  Arms: Sitagliptin 100mg qd

SUMMARY:
The aim of this combined, two part study is to evaluate the safety and glucose lowering effects of GSK256073 when administered to diabetic subjects for 12 weeks.

DETAILED DESCRIPTION:
The study will be conducted at centers in Europe and the United States. The study is being conducted in two parts. Part A (n = 90 subjects) will provide a preliminary evaluation of 12 weeks of treatment. Initiation of part B (n = 210 additional subjects) will be dependent on the results observed in part A. The emerging data from part A will be used to guide selection of the doses in Part B. Up to 8 dose levels of GSK256073 may be included in part B. The emerging exposure response relationships from the part A interim analysis will be used to guide dose selection.

Each subject enrolled in the study will undergo screening procedures, a 2 week placebo run-in period, baseline assessments, randomization, a twelve week treatment period, and a 2 week follow-up period. Following completion of the baseline visit and randomization into the study, subjects will return to the clinic for safety and efficacy assessments at Weeks 3, 6, 9, and 12. A subject's total participation in the study will last up to approximately 20 weeks. Subjects will continue their current prescribed regimen of metformin (glucophage) monotherapy and will monitor fasting blood glucose levels daily using a glucometer.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of T2DM as determined by a responsible physician based on a medical evaluation including medical history, physical examination, and laboratory tests, with onset at least 6 months prior to Screening. Subjects may be entered if they have stable hypertension or dyslipidemia on therapy. Subjects with other conditions except as noted in the Exclusion criteria may be included only if the investigator and GSK medical monitor agree that the condition is unlikely to introduce additional risk factors and will not interfere with study procedures
* HbA1c levels greater than or equal to 7.0 % and less than or equal to 9.5% at Screening
* On monotherapy with metformin at the time of screening, and at a maximum tolerated dose greater than or equal to 1000 mg for at least 2 months prior to dosing.
* Fasting plasma glucose level less than 13.3 mmol/L (240 mg/dL) at Screening
* Male or female between 20 and 70 years of age, inclusive, at the time of signing the informed consent
* Fasting Triglycerides lower than 4.52 mmol/L (400 mg/dL)
* A female subject is able to participate is she if of non-child bearing potential
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 3 days after last dose of the study medication
* Overweight with BMI greater than or equal to 25 kg/m2 for non-Asian Indians and greater than or equal to 24 kg/m2 for Asian-Indian, and less than 40 kg/m2
* The subject is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Subjects in France will be eligible only if they are affiliated to or a beneficiary of a social security category
* Subjects in other countries must meet all local and/or country-specific requirements for registration and reimbursement, as applicable

Exclusion Criteria:

* Requiring insulin therapy or use of combination oral antidiabetic medications or use of monotherapy other than metformin within the 3 months prior to screening
* Past or present disease (other than type 2 diabetes mellitus) that in the opinion of the Investigator may affect the outcome of this study
* A positive pre-study Hepatitis B surface antigen, or positive Hepatitis C result within 3 months of screening
* Renal impairment as defined by a calculated GFR less than 60 mL/min
* Any concurrent serious illness (e.g., severe COPD, history of malignancy other than skin cancer within 5 years of initial diagnosis or with evidence of recurrence) that may interfere with a subject completing the study
* Laboratory values as defined per protocol
* ECG criteria as defined per protocol
* Systolic blood pressure greater than 160 mmHg, or diastolic blood pressure greater than 100 mmHg at Screening
* History of uric acid kidney stone, and being treated with drugs for hyperuricemia including Allopurinol or Probenecid
* History of peptic ulcer disease (PUD) and/or other gastrointestinal bleeding within the 12 months prior to screening
* Use of certain blood pressure medications or certain other medications that are renally excreted as defined per protocol
* History of myopathy or CPK value greater than 3 times upper limit of normal at screening
* The subject has participated in a clinical trial and has received an investigational product within 30 days or 5 half-lives or twice the biological effect (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Any change in diet, exercise habits or smoking status within six weeks prior to screening. Any subject that cannot refrain from smoking while in the unit must be excluded
* History of sensitivity to any of the study medications, including sitagliptin or metformin, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* The subject has a positive pre-study drug screen
* History of regular alcohol consumption within 6 months of the study as defined per protocol
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Pregnant females as determined by positive serum and/or urine hCG test at screening and prior to dosing
* Lactating females
* Subjects who are unwilling or unable to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-07-13 (Actual); Primary Completion 2012-09-16 (Actual); Study Completion 2012-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (3):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miramar, Florida
- France (4):
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rueil-Malmaison
- Spain (4):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
- United Kingdom (4):
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Coventry
  - GSK Investigational Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a study in participants with Type 2 diabetes mellitus which was conducted across 14 centers in 4 countries (France [4], Spain [3], United Kingdom [4], Unites States [3]) from 13 July 2011 to 17 September 2012. Total of 89 participants were included in the pharmacokinetic population.
Groups:
- Placebo (Pooled): Eligible participants in this arm received GSK256073 matching placebo capsules twice a day (BID) and once daily orally as directed with water for 12 weeks in a fed state. According to the randomized dose regimen, participants either took 2 capsules in the morning (once daily arm) or 1 capsule each in the morning and evening (BID arms). The data for placebos-GSK256073 matched placebo BID and GSK256073 matched placebo once daily was pooled into one placebo group.
- GSK256073 5 mg BID: Eligible participants in this arm received GSK256073 5 milligrams (mg) capsules BID orally as directed with water for 12 weeks in a fed state.
- GSK256073 10 mg Once Daily: Eligible participants in this arm received GSK256073 10 mg capsules once daily orally as directed with water for 12 weeks in a fed state.
- GSK256073 25 mg BID: Eligible participants in this arm received GSK256073 25 mg capsules BID orally as directed with water for 12 weeks in a fed state.
- GSK256073 50 mg Once Daily: Eligible participants in this arm received GSK256073 50 mg capsules once daily orally as directed with water for 12 weeks in a fed state.
Period: Overall Study
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Started | 20 | 18 | 19 | 19 | 18
Completed | 18 | 17 | 16 | 14 | 17
Not Completed | 2 | 1 | 3 | 5 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo (Pooled): Eligible participants in this arm received GSK256073 matching placebo capsules BID and once daily orally as directed with water for 12 weeks in a fed state. According to the randomized dose regimen, participants either took 2 capsules in the morning (once daily arm) or 1 capsule each in the morning and evening (BID arms). The data for placebos-GSK256073 matched placebo BID and GSK256073 matched placebo once daily was pooled into one placebo group.
- GSK256073 5 mg BID: Eligible participants in this arm received GSK256073 5 mg capsules BID orally as directed with water for 12 weeks in a fed state.
- Total: Total of all reporting groups
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily | Total
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18 | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (7.01) | 60.0 (6.24) | 59.6 (8.07) | 60.2 (6.21) | 57.1 (7.30) | 58.8 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 10 | 5 | 1 | 27
  Male | 16 | 11 | 9 | 14 | 17 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 2 | 0 | 5
  White | 16 | 18 | 19 | 16 | 18 | 87
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury.
Time Frame: Up to Week 12
Population: Safety population was used which was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Participants
  Any AE | 11 | 12 | 12 | 11 | 10
  Any SAE | 1 | 0 | 0 | 2 | 0

2. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Mean of triplicate measurements at each time point was considered for the summary. Baseline was defined as pre-dose of Day 1 visit. Change from Baseline was calculated by subtracting the Baseline values from the corresponding post-treatment values. It was assessed on Baseline, Day 1 (12 hours), Day 2 (pre-dose and 12 hours), Week 3, 6 (pre-dose and 12 hours), 9 and 12.
Time Frame: Baseline (pre-dose Day 1) and up to Week 12
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Groups:
- GSK256073 5mg BID: Eligible participants in this arm received GSK256073 5 mg capsules BID orally as directed with water for 12 weeks in a fed state.
- GSK256073 10mg Once Daily: Eligible participants in this arm received GSK256073 10 mg capsules once daily orally as directed with water for 12 weeks in a fed state.
- GSK256073 25mg BID: Eligible participants in this arm received GSK256073 25 mg capsules BID orally as directed with water for 12 weeks in a fed state.
- GSK256073 50mg Once Daily: Eligible participants in this arm received GSK256073 50 mg capsules once daily orally as directed with water for 12 weeks in a fed state.
Arm/Group | Placebo (Pooled) | GSK256073 5mg BID | GSK256073 10mg Once Daily | GSK256073 25mg BID | GSK256073 50mg Once Daily
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Millimeters of mercury
  SBP, Day 1,12 hours: number analyzed (Participants) | 20 | 18 | 18 | 17 | 18
  SBP, Day 1,12 hours | 3.4 (10.48) | 0.9 (10.73) | 4.9 (19.88) | 3.0 (12.90) | 1.9 (11.04)
  SBP, Day 2, pre-dose: number analyzed (Participants) | 20 | 18 | 18 | 18 | 18
  SBP, Day 2, pre-dose | -0.8 (10.66) | -6.5 (11.30) | -7.7 (10.97) | -1.7 (7.73) | -4.7 (9.25)
  SBP, Day 2, 12 hours: number analyzed (Participants) | 20 | 17 | 18 | 18 | 18
  SBP, Day 2, 12 hours | 0.7 (11.84) | -3.8 (8.34) | 1.1 (11.76) | 1.7 (7.86) | -1.8 (11.16)
  SBP, Week 3: number analyzed (Participants) | 20 | 17 | 17 | 18 | 18
  SBP, Week 3 | 3.7 (13.68) | -3.9 (11.83) | 0.5 (12.41) | -1.7 (10.71) | -1.1 (8.78)
  SBP, Day 6, pre-dose: number analyzed (Participants) | 19 | 17 | 17 | 17 | 18
  SBP, Day 6, pre-dose | -0.1 (11.26) | -7.7 (12.96) | -3.4 (9.07) | -5.3 (16.93) | -5.8 (8.19)
  SBP, Day 6, 12 hours: number analyzed (Participants) | 19 | 17 | 17 | 16 | 18
  SBP, Day 6, 12 hours | 6.6 (15.32) | -2.5 (14.05) | 1.0 (10.83) | 2.7 (12.76) | 1.6 (7.51)
  SBP, Week 9: number analyzed (Participants) | 19 | 17 | 16 | 16 | 17
  SBP, Week 9 | 4.0 (11.93) | -9.1 (14.02) | -1.6 (10.27) | -2.0 (11.73) | -3.8 (10.57)
  SBP, Week 12: number analyzed (Participants) | 18 | 17 | 16 | 15 | 17
  SBP, Week 12 | 2.3 (9.85) | -6.4 (8.08) | -0.3 (7.95) | 2.8 (13.13) | 0.4 (10.59)
  DBP, Day 1,12 hours: number analyzed (Participants) | 20 | 18 | 18 | 17 | 18
  DBP, Day 1,12 hours | 1.4 (6.66) | 0.6 (7.42) | 2.0 (6.00) | -0.5 (7.69) | 3.2 (8.55)
  DBP, Day 2, pre-dose: number analyzed (Participants) | 20 | 18 | 18 | 18 | 18
  DBP, Day 2, pre-dose | -1.2 (6.89) | -2.1 (7.46) | -2.1 (5.27) | -1.7 (5.15) | -0.2 (6.37)
  DBP, Day 2, 12 hours: number analyzed (Participants) | 20 | 17 | 18 | 18 | 18
  DBP, Day 2, 12 hours | 0.8 (6.17) | -0.6 (6.57) | 1.4 (4.89) | 0.8 (5.65) | 2.0 (6.62)
  DBP, Week 3: number analyzed (Participants) | 20 | 17 | 17 | 18 | 18
  DBP, Week 3 | 2.2 (6.59) | 0.3 (5.32) | -0.1 (8.42) | -0.5 (6.75) | 1.0 (6.43)
  DBP, Day 6, pre-dose: number analyzed (Participants) | 19 | 17 | 17 | 17 | 18
  DBP, Day 6, pre-dose | 1.3 (6.74) | -4.7 (8.96) | -0.4 (6.82) | -2.0 (9.56) | -1.4 (4.73)
  DBP, Day 6, 12 hours: number analyzed (Participants) | 19 | 17 | 17 | 16 | 18
  DBP, Day 6, 12 hours | 2.9 (7.94) | -1.7 (8.01) | 1.0 (5.55) | 0.6 (5.80) | 1.5 (7.37)
  DBP, Week 9: number analyzed (Participants) | 19 | 17 | 16 | 16 | 17
  DBP, Week 9 | 3.3 (7.63) | -2.8 (8.79) | 0.1 (7.66) | -0.9 (8.23) | -1.2 (7.65)
  DBP, Week 12: number analyzed (Participants) | 18 | 17 | 16 | 15 | 17
  DBP, Week 12 | 0.1 (5.95) | -3.4 (8.69) | 0.7 (6.51) | 0.9 (7.03) | 0.3 (6.30)

3. Primary Outcome: Change From Baseline in Heart Rate
Description: Mean of triplicate measurements at each time point was considered for the summary. Baseline was defined as pre-dose of Day 1 visit. Change from Baseline was calculated by subtracting the Baseline values from the corresponding post-treatment values. It was assessed on Baseline (pre-dose Day 1), Day 1 (12 hours), Day 2, Week 3, 6, 9 and 12.
Time Frame: Baseline (pre-dose Day 1) and up to Week 12
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo (Pooled) | GSK256073 5mg BID | GSK256073 10mg Once Daily | GSK256073 25mg BID | GSK256073 50mg Once Daily
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Beats per minute
  Day 1,12 hours: number analyzed (Participants) | 20 | 18 | 18 | 18 | 18
  Day 1,12 hours | 2.5 (5.39) | -1.0 (4.64) | 1.1 (7.77) | 1.3 (7.07) | 0.7 (7.93)
  Day 2, pre-dose: number analyzed (Participants) | 20 | 18 | 18 | 18 | 18
  Day 2, pre-dose | 1.2 (4.79) | 1.2 (6.93) | 2.6 (5.01) | 0.9 (6.99) | 1.3 (7.74)
  Day 2, 12 hours: number analyzed (Participants) | 20 | 17 | 18 | 18 | 18
  Day 2, 12 hours | 3.3 (6.80) | 1.9 (6.81) | 4.6 (7.02) | 3.8 (7.62) | 1.5 (7.71)
  Week 3: number analyzed (Participants) | 20 | 17 | 17 | 18 | 18
  Week 3 | 3.2 (5.44) | 1.2 (8.41) | 3.1 (7.47) | 0.1 (4.81) | 1.2 (7.95)
  Day 6, pre-dose: number analyzed (Participants) | 19 | 17 | 17 | 17 | 18
  Day 6, pre-dose | -0.9 (6.53) | -1.6 (7.62) | 0.5 (6.89) | 3.1 (14.29) | -1.2 (9.88)
  Day 6, 12 hours: number analyzed (Participants) | 19 | 17 | 17 | 16 | 18
  Day 6, 12 hours | 2.9 (6.56) | 2.2 (9.13) | 3.3 (7.48) | 6.6 (11.16) | -3.8 (9.14)
  Week 9: number analyzed (Participants) | 19 | 17 | 16 | 16 | 17
  Week 9 | 1.7 (6.44) | 3.6 (8.71) | 4.9 (11.40) | 4.4 (9.26) | 3.2 (9.10)
  Week 12: number analyzed (Participants) | 18 | 17 | 16 | 15 | 17
  Week 12 | 2.8 (6.95) | 1.1 (10.59) | 4.1 (10.12) | 3.9 (9.98) | -0.5 (8.46)

4. Primary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs) Findings
Description: Single 12-lead ECGs were obtained at each time point during the study using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and QTc intervals. It was assessed at Baseline (pre-dose Day 1), Day 2, Week 3, Week 6 and 12. Participants with normal, abnormal not clinically significant and abnormal clinically significant ECG were presented.
Time Frame: Up to Week 20
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Participants
  Day 1: normal | 12 | 14 | 13 | 18 | 12
  Day 1: abnormal not clinically significant | 8 | 4 | 6 | 1 | 6
  Day 1: abnormal clinically significant | 0 | 0 | 0 | 0 | 0
  Day 2: number analyzed (Participants) | 20 | 17 | 18 | 17 | 18
  Day 2: normal | 14 | 14 | 13 | 16 | 12
  Day 2: abnormal not clinically significant | 6 | 3 | 5 | 1 | 6
  Day 2: abnormal clinically significant | 0 | 0 | 0 | 0 | 0
  Week 3: number analyzed (Participants) | 20 | 17 | 16 | 18 | 17
  Week 3: normal | 17 | 14 | 13 | 16 | 13
  Week 3: abnormal not clinically significant | 3 | 3 | 3 | 2 | 4
  Week 3: abnormal clinically significant | 0 | 0 | 0 | 0 | 0
  Week 6: number analyzed (Participants) | 19 | 17 | 17 | 17 | 18
  Week 6: normal | 16 | 14 | 14 | 12 | 12
  Week 6: abnormal not clinically significant | 3 | 3 | 3 | 4 | 6
  Week 6: abnormal clinically significant | 0 | 0 | 0 | 1 | 0
  Week 12: number analyzed (Participants) | 18 | 17 | 16 | 15 | 17
  Week 12: normal | 10 | 14 | 13 | 12 | 14
  Week 12: abnormal not clinically significant | 8 | 3 | 3 | 3 | 3
  Week 12: abnormal clinically significant | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinical Chemistry Abnormalities of Potential Clinical Importance (PCI)
Description: Clinical chemistry parameters included blood urea nitrogen (BUN), potassium, aspartate aminotransferase (AST), total bilirubin, direct bilirubin, creatinine, chloride, alanine aminotransferase (ALT), uric acid, fasting glucose, total carbon dioxide, gamma glutamyltransferase (GGT), albumin, sodium, calcium, alkaline phosphatase (ALP), total protein, creatine phosphokinase (CPK) and fasting lipid panel including total cholesterol, triglycerides, high density lipoprotein (HDL) cholesterol and low density lipoprotein (LDL) cholesterol. It was assessed on Baseline (pre-dose Day 1), Week 3 and 12. Data for parameters with high and low of PCI is provided.
Time Frame: Up to Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- GSK256073 50 mg Once Daily: Eligible participants in this arm received GSK256073 25 mg capsules BID orally as directed with water for 12 weeks in a fed state.
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Participants
  Potassium, high | 1 | 0 | 1 | 0 | 1
  Potassium, low | 1 | 0 | 0 | 0 | 0
  Albumin, low | 2 | 0 | 0 | 0 | 0
  Creatine kinase, high | 2 | 1 | 1 | 0 | 0
  Creatinine, high | 1 | 0 | 0 | 0 | 0
  Total bilirubin, high | 0 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Hematology Abnormalities of Potential Clinical Importance (PCI)
Description: Hematology parameters included platelet, red blood cell (RBC) count, mean corpuscular volume (MCV), neutrophils, white blood cell (WBC) count (absolute), mean corpuscular hemoglobin (MCH), lymphocytes, reticulocyte count, mean corpuscular hemoglobin concentration (MCHC), monocytes, hemoglobin, eosinophils, hematocrit and basophils. It was assessed on Baseline (pre-dose Day 1) and 12. Data for parameters with high and low of PCI is provided.
Time Frame: Up to Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Participants
  Total neutrophils, low | 3 | 0 | 0 | 1 | 0
  Platelet count, low | 1 | 1 | 0 | 0 | 1
  Lymphocytes, low | 0 | 0 | 0 | 2 | 0
  WBC, low | 0 | 0 | 0 | 1 | 0

7. Primary Outcome: Number of Participants With Abnormal Urinalysis: Glucose, Protein, Blood and Ketones by Dipstick
Description: Urinalysis parameters included glucose, protein, blood and ketones by dipstick. It was assessed on Baseline (Day -1) and 12. Urine glucose was measured as grams per deciliter (G/dL).
Time Frame: Up to Week 12
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Participants
  Urine glucose, Day -1, Negative: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine glucose, Day -1, Negative | 13 | 11 | 14 | 10 | 14
  Urine glucose, Day -1, Trace: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine glucose, Day -1, Trace | 0 | 0 | 0 | 2 | 0
  Urine glucose, Day -1, Trace or 1/10 g/dL: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine glucose, Day -1, Trace or 1/10 g/dL | 1 | 4 | 2 | 3 | 1
  Urine glucose, Day -1, 1+ or 1/4 g/dL: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine glucose, Day -1, 1+ or 1/4 g/dL | 2 | 1 | 2 | 3 | 2
  Urine glucose, Day -1, 2+ or 1/2 g/dL: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine glucose, Day -1, 2+ or 1/2 g/dL | 0 | 1 | 1 | 0 | 0
  Urine glucose, Day -1, 3+ or 1 g/dL: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine glucose, Day -1, 3+ or 1 g/dL | 3 | 1 | 0 | 1 | 1
  Urine glucose, Day 41, Negative: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine glucose, Day 41, Negative | 13 | 12 | 13 | 12 | 13
  Urine glucose, Day 41, Trace: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine glucose, Day 41, Trace | 1 | 0 | 0 | 0 | 0
  Urine glucose, Day 41, Trace or 1/10 g/dL: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine glucose, Day 41, Trace or 1/10 g/dL | 1 | 3 | 1 | 1 | 2
  Urine glucose, Day 41, 1+ or 1/4 g/dL: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine glucose, Day 41, 1+ or 1/4 g/dL | 1 | 0 | 2 | 1 | 1
  Urine glucose, Day 41, 2+ or 1/2 g/dL: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine glucose, Day 41, 2+ or 1/2 g/dL | 0 | 0 | 0 | 1 | 0
  Urine glucose, Day 41, 3+ or 1 g/dL: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine glucose, Day 41, 3+ or 1 g/dL | 3 | 2 | 0 | 2 | 1
  Urine glucose, Week 12, Negative: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine glucose, Week 12, Negative | 13 | 13 | 13 | 8 | 15
  Urine glucose, Week 12, Trace: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine glucose, Week 12, Trace | 0 | 0 | 0 | 1 | 0
  Urine glucose, Week 12, Trace or 1/10 g/dL: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine glucose, Week 12, Trace or 1/10 g/dL | 1 | 2 | 0 | 1 | 0
  Urine glucose, Week 12, 1+ or 1/4 g/dL: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine glucose, Week 12, 1+ or 1/4 g/dL | 2 | 1 | 0 | 3 | 0
  Urine glucose, Week 12, 2+ or 1/2 g/dL: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine glucose, Week 12, 2+ or 1/2 g/dL | 1 | 0 | 1 | 0 | 0
  Urine glucose, Week 12, 3+ or 1 g/dL: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine glucose, Week 12, 3+ or 1 g/dL | 1 | 1 | 1 | 1 | 1
  Urine ketones, Day -1, Negative: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine ketones, Day -1, Negative | 18 | 17 | 19 | 18 | 17
  Urine ketones, Day -1, Trace: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine ketones, Day -1, Trace | 1 | 0 | 0 | 1 | 1
  Urine ketones, Day -1, 1+: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine ketones, Day -1, 1+ | 0 | 1 | 0 | 0 | 0
  Urine ketones, Day -1, 2+: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Urine ketones, Day 41, Negative: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine ketones, Day 41, Negative | 18 | 15 | 13 | 14 | 14
  Urine ketones, Day 41, Trace: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine ketones, Day 41, Trace | 1 | 1 | 2 | 2 | 3
  Urine ketones, Day 41, 1+ or 1/4: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine ketones, Day 41, 1+ or 1/4 | 0 | 0 | 1 | 1 | 0
  Urine ketones, Day 41, 2+: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine ketones, Day 41, 2+ | 0 | 1 | 0 | 0 | 0
  Urine ketones, Week 12, Negative: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine ketones, Week 12, Negative | 17 | 14 | 15 | 12 | 12
  Urine ketones, Week 12, Trace: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine ketones, Week 12, Trace | 1 | 3 | 0 | 1 | 3
  Urine ketones, Week 12, 1+ or 1/4: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine ketones, Week 12, 1+ or 1/4 | 0 | 0 | 0 | 1 | 1
  Urine ketones, Week 12, 2+: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Urine occult blood, Day -1, Negative: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine occult blood, Day -1, Negative | 18 | 17 | 16 | 17 | 18
  Urine occult blood, Day -1, Trace: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine occult blood, Day -1, Trace | 1 | 0 | 3 | 0 | 0
  Urine occult blood, Day -1, 1+: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine occult blood, Day -1, 1+ | 0 | 1 | 0 | 2 | 0
  Urine occult blood, Day 41, Negative: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine occult blood, Day 41, Negative | 19 | 15 | 15 | 15 | 17
  Urine occult blood, Day 41, Trace: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine occult blood, Day 41, Trace | 0 | 2 | 1 | 2 | 0
  Urine occult blood, Day 41, 1+: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Urine occult blood, Week 12, Negative: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine occult blood, Week 12, Negative | 17 | 15 | 15 | 12 | 16
  Urine occult blood, Week 12, Trace: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine occult blood, Week 12, Trace | 0 | 0 | 0 | 1 | 0
  Urine occult blood, Week 12, 1+: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine occult blood, Week 12, 1+ | 1 | 2 | 0 | 1 | 0
  Urine protein, Day -1, Negative: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine protein, Day -1, Negative | 18 | 13 | 12 | 14 | 14
  Urine protein, Day -1, Trace: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine protein, Day -1, Trace | 0 | 2 | 4 | 2 | 4
  Urine protein, Day -1, 1+: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine protein, Day -1, 1+ | 0 | 2 | 2 | 2 | 0
  Urine protein, Day -1, 2+: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine protein, Day -1, 2+ | 1 | 1 | 1 | 0 | 0
  Urine protein, Day -1, 3+: number analyzed (Participants) | 19 | 18 | 19 | 19 | 18
  Urine protein, Day -1, 3+ | 0 | 0 | 0 | 1 | 0
  Urine protein, Day 41, Negative: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine protein, Day 41, Negative | 17 | 12 | 13 | 15 | 14
  Urine protein, Day 41, Trace: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine protein, Day 41, Trace | 1 | 3 | 1 | 0 | 3
  Urine protein, Day 41, 1+: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine protein, Day 41, 1+ | 1 | 1 | 1 | 1 | 0
  Urine protein, Day 41, 2+: number analyzed (Participants) | 19 | 17 | 16 | 17 | 17
  Urine protein, Day 41, 2+ | 0 | 1 | 1 | 1 | 0
  Urine protein, Day 41, 3+: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Urine protein, Week 12, Negative: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine protein, Week 12, Negative | 15 | 12 | 14 | 9 | 14
  Urine protein, Week 12, Trace: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine protein, Week 12, Trace | 2 | 2 | 0 | 3 | 2
  Urine protein, Week 12, 1+: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine protein, Week 12, 1+ | 1 | 2 | 1 | 1 | 0
  Urine protein, Week 12, 2+: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine protein, Week 12, 2+ | 0 | 1 | 0 | 0 | 0
  Urine protein, Week 12, 3+: number analyzed (Participants) | 18 | 17 | 15 | 14 | 16
  Urine protein, Week 12, 3+ | 0 | 0 | 0 | 1 | 0

8. Primary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 12
Description: Blood samples for analysis of HbA1c were collected at Baseline (Day -1), Day 41, Week 9 and Week 12. Change from Baseline was calculated by subtracting the Baseline values from the corresponding post-treatment values. Baseline was defined as Day -1 visit. Statistics is provided for least square mean at Week 12.
Time Frame: Baseline (Day -1) and up to Week 12
Population: Pharmacodynamic (PD) population comprised of all participants who provide pharmacodynamic data. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of Glycosylated Hemoglobin
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Percentage of Glycosylated Hemoglobin
  Day 41: number analyzed (Participants) | 19 | 17 | 17 | 17 | 18
  Day 41 | -0.34 (0.709) | -0.18 (0.555) | -0.37 (0.443) | -0.42 (0.423) | -0.44 (0.370)
  Week 9: number analyzed (Participants) | 18 | 17 | 16 | 16 | 17
  Week 9 | -0.44 (0.808) | -0.24 (0.608) | -0.48 (0.503) | -0.56 (0.512) | -0.59 (0.464)
  Week 12: number analyzed (Participants) | 18 | 17 | 16 | 15 | 17
  Week 12 | -0.36 (0.698) | -0.14 (0.778) | -0.46 (0.507) | -0.56 (0.562) | -0.64 (0.630)
Statistical Analysis 1: Comparison: Placebo (Pooled) vs GSK256073 5 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.24, 95% CI 2-sided [-0.13 to 0.60]
Statistical Analysis 2: Comparison: Placebo (Pooled) vs GSK256073 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.37 to 0.35]
Statistical Analysis 3: Comparison: Placebo (Pooled) vs GSK256073 25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.49 to 0.23]
Statistical Analysis 4: Comparison: Placebo (Pooled) vs GSK256073 50 mg Once Daily; Test type: Superiority or Other; Mean Difference (Net) = -0.30, 95% CI 2-sided [-0.66 to 0.06]

9. Secondary Outcome: Change From Baseline in 12 Hour Non-esterified Fatty Acids (NEFA) and Glucose Weighted Mean Concentration Value at Day 2 and at Week 6
Description: Change from Baseline was calculated by subtracting the Baseline values from the corresponding post-treatment values. Baseline was defined as weighted mean value at Day 1 visit. Statistics is provided for least square mean at Week 6. It was assessed on Baseline (Day 1), Day 2 and Week 6.
Time Frame: Baseline (Day 1) and up to Week 6
Population: PD population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Groups:
- GSK256073 10 mg qd: Eligible participants in this arm received GSK256073 10 mg capsules once daily orally as directed with water for 12 weeks in a fed state.
- GSK256073 50 mg qd: Eligible participants in this arm received GSK256073 50 mg capsules once daily orally as directed with water for 12 weeks in a fed state.
Arm/Group | Placebo (Pooled) | GSK256073 5 mg Bid | GSK256073 10 mg qd | GSK256073 25 mg Bid | GSK256073 50 mg qd
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Millimoles per liter
  Glucose, Day 2: number analyzed (Participants) | 20 | 17 | 18 | 18 | 18
  Glucose, Day 2 | 0.462 (1.0525) | -0.502 (2.0948) | 0.036 (1.0464) | -0.517 (0.8577) | -0.076 (0.9745)
  Glucose, Week 6: number analyzed (Participants) | 19 | 17 | 17 | 16 | 18
  Glucose, Week 6 | 0.009 (1.8099) | -0.786 (3.1101) | -0.502 (1.2995) | -0.647 (1.0043) | -0.544 (1.3403)
  NEFA, Day 2: number analyzed (Participants) | 20 | 17 | 18 | 18 | 18
  NEFA, Day 2 | -0.0152 (0.08082) | -0.1307 (0.09016) | -0.1326 (0.12437) | -0.1926 (0.13820) | -0.1503 (0.09720)
  NEFA, Week 6: number analyzed (Participants) | 19 | 17 | 17 | 16 | 18
  NEFA, Week 6 | -0.0457 (0.07154) | -0.0342 (0.17352) | -0.0423 (0.08431) | -0.0293 (0.22736) | -0.1032 (0.11673)
Statistical Analysis 1: Comparison: Placebo (Pooled) vs GSK256073 5 mg Bid; Test type: Superiority or Other; Mean Difference (Net) = -0.551, 95% CI 2-sided [-1.645 to 0.543] — Comparison for glucose
Statistical Analysis 2: Comparison: Placebo (Pooled) vs GSK256073 10 mg qd; Test type: Superiority or Other; Mean Difference (Net) = -0.382, 95% CI 2-sided [-1.472 to 0.708] — Comparison for glucose
Statistical Analysis 3: Comparison: Placebo (Pooled) vs GSK256073 25 mg Bid; Test type: Superiority or Other; Mean Difference (Net) = -0.590, 95% CI 2-sided [-1.696 to 0.516] — Comparison for glucose
Statistical Analysis 4: Comparison: Placebo (Pooled) vs GSK256073 50 mg qd; Test type: Superiority or Other; Mean Difference (Net) = -0.595, 95% CI 2-sided [-1.669 to 0.480] — Comparison for glucose
Statistical Analysis 5: Comparison: Placebo (Pooled) vs GSK256073 5 mg Bid; Test type: Superiority or Other; Mean Difference (Net) = 0.036, 95% CI 2-sided [-0.042 to 0.113] — Comparison for NEFA
Statistical Analysis 6: Comparison: Placebo (Pooled) vs GSK256073 10 mg qd; Test type: Superiority or Other; Mean Difference (Net) = 0.004, 95% CI 2-sided [-0.073 to 0.081] — Comparison for NEFA
Statistical Analysis 7: Comparison: Placebo (Pooled) vs GSK256073 25 mg Bid; Test type: Superiority or Other; Mean Difference (Net) = 0.021, 95% CI 2-sided [-0.058 to 0.099] — Comparison for NEFA
Statistical Analysis 8: Comparison: Placebo (Pooled) vs GSK256073 50 mg qd; Test type: Superiority or Other; Mean Difference (Net) = -0.083, 95% CI 2-sided [-0.160 to -0.007] — Comparison for NEFA

10. Secondary Outcome: GSK256073 AUC and HbA1c at Week 12 Was Evaluated to Establish the Exposure-response Pharmacokinetic/Pharmacodynamic (PK/PD) Relationship
Description: The relationships between drug exposure and HbA1c and relative PD endpoints of interest was planned to be plotted graphically. The data for this outcome measure was not collected.
Time Frame: Up to Week 12
Population: PD population. The data for this outcome measure was not collected.
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 12
Description: Mean of triplicate measurements at pre-dose time point were considered for the summary. Change from Baseline was calculated by subtracting the Baseline values from the corresponding post-treatment values. Baseline was defined as mean of Day 1 pre-dose visit. Statistics is provided for least square mean at Week 12. It was assessed on Day 1 (pre-dose), 2 (pre-dose), Week 6 (pre-dose) and Week 12.
Time Frame: Baseline (Day 1) and up to Week 12
Population: PD population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Millimoles per liter
  Day 2: number analyzed (Participants) | 20 | 16 | 18 | 18 | 18
  Day 2 | 0.09 (0.723) | -0.05 (1.186) | 0.04 (1.019) | 0.04 (1.611) | -0.34 (0.590)
  Week 6: number analyzed (Participants) | 19 | 17 | 17 | 17 | 18
  Week 6 | -0.25 (1.933) | -0.82 (2.910) | -1.06 (1.472) | -0.62 (1.289) | -0.91 (1.030)
  Week 12: number analyzed (Participants) | 18 | 17 | 16 | 15 | 17
  Week 12 | -0.64 (1.439) | -0.85 (2.547) | -0.71 (1.290) | -0.44 (0.913) | -0.83 (1.497)
Statistical Analysis 1: Comparison: Placebo (Pooled) vs GSK256073 5 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.79 to 0.94]
Statistical Analysis 2: Comparison: Placebo (Pooled) vs GSK256073 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.90 to 0.82]
Statistical Analysis 3: Comparison: Placebo (Pooled) vs GSK256073 25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.90 to 0.85]
Statistical Analysis 4: Comparison: Placebo (Pooled) vs GSK256073 50 mg Once Daily; Test type: Superiority or Other; Mean Difference (Net) = -0.42, 95% CI 2-sided [-1.27 to 0.42]

12. Secondary Outcome: Change From Baseline in Fasting Insulin at Week 12
Description: as for outcome 11
Time Frame: Baseline (Day 1) and up to Week 12
Population: PD population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomoles per liter
Groups:
- GSK256073 50 mg qd: Eligible participants in this arm received GSK256073 25 mg capsules BID orally as directed with water for 12 weeks in a fed state.
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg qd | GSK256073 25 mg BID | GSK256073 50 mg qd
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Picomoles per liter
  Day 2: number analyzed (Participants) | 20 | 16 | 18 | 18 | 18
  Day 2 | -1.1 (73.81) | 19.1 (52.10) | 6.6 (34.90) | -2.8 (26.41) | 0.2 (22.75)
  Week 6: number analyzed (Participants) | 19 | 17 | 17 | 17 | 18
  Week 6 | -3.9 (25.74) | -9.1 (38.84) | 2.9 (20.77) | -6.0 (50.97) | 2.6 (78.83)
  Week 12: number analyzed (Participants) | 14 | 14 | 15 | 13 | 15
  Week 12 | 27.3 (139.30) | 14.7 (38.66) | -2.0 (25.80) | 33.4 (80.94) | 4.7 (43.42)
Statistical Analysis 1: Comparison: Placebo (Pooled) vs GSK256073 5 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 2.27, 95% CI 2-sided [-48.62 to 53.16]
Statistical Analysis 2: Comparison: Placebo (Pooled) vs GSK256073 10 mg qd; Test type: Superiority or Other; Mean Difference (Net) = -7.67, 95% CI 2-sided [-58.04 to 42.70]
Statistical Analysis 3: Comparison: Placebo (Pooled) vs GSK256073 25 mg BID; Test type: Superiority or Other; Median Difference (Net) = 24.08, 95% CI 2-sided [-27.75 to 75.92]
Statistical Analysis 4: Comparison: Placebo (Pooled) vs GSK256073 50 mg qd; Test type: Superiority or Other; Mean Difference (Net) = -2.09, 95% CI 2-sided [-52.72 to 48.53]

13. Secondary Outcome: Summary of Homeostatic Model Assessment (HOMA) Index Calculated From Change From Baseline in Fasting Insulin and Fasting Glucose at Week 12
Description: Mean of triplicate measurements at pre-dose time point was considered for the summary. HOMA was calculated by multiplying insulin concentration with glucose concentration divided by 22.5. Change from Baseline for insulin and glucose was calculated by subtracting the Baseline values from the corresponding post-treatment values. Baseline was defined as mean of Day 1 pre-dose visit. Statistics is provided for least square mean. It was assessed on Day 1 (pre-dose), 2 (pre-dose), Week 6 (pre-dose) and Week 12.
Time Frame: Baseline (Day 1) and up to Week 12
Population: PD population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Index
  Day 2: number analyzed (Participants) | 20 | 16 | 18 | 18 | 18
  Day 2 | 0.2 (4.24) | 1.1 (3.83) | 0.3 (1.98) | -0.2 (1.73) | -0.2 (1.33)
  Week 6: number analyzed (Participants) | 19 | 17 | 17 | 17 | 18
  Week 6 | -0.6 (3.13) | -1.4 (4.11) | -0.3 (1.75) | -0.4 (3.46) | -0.7 (3.76)
  Week 12: number analyzed (Participants) | 14 | 14 | 15 | 13 | 15
  Week 12 | -0.0 (3.57) | 0.0 (2.47) | -0.3 (2.08) | 1.5 (4.17) | -0.1 (3.44)

14. Secondary Outcome: Change From Baseline in Fructosamine at Week 6 and Week 12
Description: Change from Baseline was calculated by subtracting the Baseline values from the corresponding post-treatment values. Baseline was defined as mean of Day -1 visit. Statistics is provided for least square mean. It was assessed on Baseline (Day -1), Day 41 and Week 12.
Time Frame: Baseline (Day -1) and Week 12
Population: PD population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Number analyzed (Participants) | 20 | 18 | 19 | 19 | 18
Micromoles per liter
  Day 41: number analyzed (Participants) | 19 | 17 | 16 | 15 | 16
  Day 41 | -14.9 (33.59) | -18.8 (34.49) | -21.2 (24.51) | -26.3 (25.73) | -21.1 (26.39)
  Week 12: number analyzed (Participants) | 18 | 17 | 15 | 14 | 17
  Week 12 | -22.3 (27.92) | -16.4 (37.43) | -30.7 (21.71) | -25.4 (33.74) | -36.1 (37.23)
Statistical Analysis 1: Comparison: Placebo (Pooled) vs GSK256073 5 mg BID; Test type: Superiority or Other; Mean Difference (Net) = -1.58, 95% CI 2-sided [-19.36 to 16.20]
Statistical Analysis 2: Comparison: Placebo (Pooled) vs GSK256073 10 mg Once Daily; Test type: Superiority or Other; Mean Difference (Net) = -15.10, 95% CI 2-sided [-33.00 to 2.81]
Statistical Analysis 3: Comparison: Placebo (Pooled) vs GSK256073 25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = -14.09, 95% CI 2-sided [-32.41 to 4.23]
Statistical Analysis 4: Comparison: Placebo (Pooled) vs GSK256073 50 mg Once Daily; Test type: Superiority or Other; Mean Difference (Net) = -19.12, 95% CI 2-sided [-36.55 to -1.68]

15. Secondary Outcome: Number of Participants With HbA1c < 7.0% and < 6.5%
Description: Data has been presented for number of participants with their corresponding percentages with HbA1c <7.0% and <6.5%.
Time Frame: Up to Week 12
Population: PD population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
Number analyzed (Participants) | 18 | 17 | 16 | 15 | 17
Participants
  <7% | 4 | 3 | 2 | 3 | 11
  <6.5% | 2 | 0 | 0 | 1 | 4

ADVERSE EVENTS:
Time Frame: Up to Week 12.
Description: Safety population used for assessment of safety results.
Arm/Group | Placebo (Pooled) | GSK256073 5 mg BID | GSK256073 10 mg Once Daily | GSK256073 25 mg BID | GSK256073 50 mg Once Daily
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18 | 0/19 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/18 | 0/19 | 2/19 | 0/18
Other Adverse Events (participants affected / at risk) | 11/20 | 12/18 | 12/19 | 10/19 | 10/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Pooled) (N=20) | GSK256073 5 mg BID (N=18) | GSK256073 10 mg Once Daily (N=19) | GSK256073 25 mg BID (N=19) | GSK256073 50 mg Once Daily (N=18)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Pooled) (N=20) | GSK256073 5 mg BID (N=18) | GSK256073 10 mg Once Daily (N=19) | GSK256073 25 mg BID (N=19) | GSK256073 50 mg Once Daily (N=18)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Blood uric acid decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contrast media reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.